CLINICAL TRIAL: NCT03072966
Title: Development of Distress Management Algorithms Using Mobile Device Based Health Logs in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Il Yong Chung, Clinical Assistant Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S2016-1188-0004
Record Dates: First submitted 2017-02-23; First posted 2017-03-08 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Quality of Life
Keywords: Distress; Exercise; Wearable device; Smartphone
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Distress screening group (Experimental): Physical activities will be monitored by wearable device. Patient-reported outcomes including distress, depression, physical activities and quality of life are going to be collected by questionnaires based on smartphone application and paper. The algorithm of distress screening will be developed with the analysis of patterns of physical activities.
  Interventions: Device: Wearable device (Fitbit Charge HR® or Fitbit Alta ®)

INTERVENTIONS:
Device: Wearable device (Fitbit Charge HR® or Fitbit Alta ®) — Physical activities will be monitored by wearable device.

SUMMARY:
Distress monitoring is an important issue in cancer survivors. However, conventional distress screening is very difficult to perform. This study investigates the efficacy of wearable device as a tool of distress monitoring in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Stage 0-III breast cancer

Exclusion Criteria:

* Stage IV breast cancer
* Breast cancer recurrence or metastasis
* Severe medical illness

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of distress screening of wearable device | 6months
  The results of distress screening questionnaire and patterns of physical activities are going to be compared. The association between those two data will be analyzed. Using data of physical activities, the prediction model of distress will be tested and validated.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jung M, Lee S, Kim J, Kim H, Ko B, Son BH, Ahn SH, Park YR, Cho D, Chung H, Park HJ, Lee M, Lee JW, Chung S, Chung IY. A Mobile Technology for Collecting Patient-Reported Physical Activity and Distress Outcomes: Cross-Sectional Cohort Study. JMIR Mhealth Uhealth. 2020 May 4;8(5):e17320. doi: 10.2196/17320. PMID 32364508
- [Derived] Chung IY, Jung M, Park YR, Cho D, Chung H, Min YH, Park HJ, Lee M, Lee SB, Chung S, Son BH, Ahn SH, Lee JW. Exercise Promotion and Distress Reduction Using a Mobile App-Based Community in Breast Cancer Survivors. Front Oncol. 2020 Jan 10;9:1505. doi: 10.3389/fonc.2019.01505. eCollection 2019. PMID 31998651
- [Derived] Chung IY, Jung M, Lee SB, Lee JW, Park YR, Cho D, Chung H, Youn S, Min YH, Park HJ, Lee M, Chung S, Son BH, Ahn SH. An Assessment of Physical Activity Data Collected via a Smartphone App and a Smart Band in Breast Cancer Survivors: Observational Study. J Med Internet Res. 2019 Sep 6;21(9):13463. doi: 10.2196/13463. PMID 31493319